CLINICAL TRIAL: NCT04695860
Title: An Investigator-sponsored Phase 3b Open-label Study of Anti- FGF23 Antibody Burosumab (KRN23) in Adult Patients With Xlinked Hypophosphatemia (XLH) in GERmany - BurGER
Brief Title: Anti-FGF23 (Burosumab) in Adult Patients With XLH
Acronym: BurGER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUR03
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: X-linked Hypophosphatemia
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label Burosumab (Experimental): Burosumab Q4W, 1mg/kg body weight s.c.
  Interventions: Drug: Burosumab

INTERVENTIONS:
Drug: Burosumab — Q4w, 1mg/kg Body weight, s.c.

SUMMARY:
X-linked hypophosphatemia (XLH) rare genetic disorder due by inactivating mutations in the PHEX gene leading to increased levels in FGF-23. Elevated FGF-23 reduces renal phosphate reabsorbtion and and limits 1-alpha hydroxylase driven Vitamin D activation, eventually leading to phosphate wasting, defective bone mineralization and additional health issues.

Burosumab is a recombinant fully human IgG1 monoclonal antibody developed to treat XLH by binding FGF23, thereby restoring normal phosphate homeostasis.

BUR03 is a Phase 3b open-label, single-arm, single-center study to confirm the efficacy and safety of Burosumab treatment in adult (age ≥18 years) XLH patients without upper age limit and irrespective of baseline pain level and to further evaluate the efficacy in this cohort and the assocaited effect of treatment on physical functioning, mobility and activity.

The study aims at enrolling and treating 34 subjects with a confirmed diagnosis of XLH with q4w s.c. injection of Burosumab 1mg/kg body weight over 48 weeks.

Primary objective is to attiain normal serum phosphorus levels, secondary objectives include key parameters of physical function and activity, mobility and mineral homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years, inclusive
* Diagnosis of X-linked Hypophosphatemia supported by classic clinical features of adult XLH (e.g. short statue or bowed legs, clinical symptoms as judged by the investigator) and at least one of the following at Screening visit:

  * documented PHEX mutation in either the patient, or
  * in a directly related family member with appropriate X-linked inheritance
  * Increased serum levels of c-term FGF23 or iFGF23
* Biochemical findings consistent with XLH at Screening visit following overnight fasting:

  * Serum phosphorus level or
  * TmP/GFR below lab specific lower limit of normal (LLN)
* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min (using the Chronic Kidney Disease Epidemiology Collaboration equitation) or eGFR of 30 up to 60 mL/min at Screening visit with confirmation that the renal insufficiency is not due to nephrocalcinosis
* Subjects who provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures.
* Participants must, in the opinion of the investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments.
* Females of child-bearing potential must have a negative urine pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not to be of child-bearing potential include those who have been in menopause for at least 2 years prior to Screening, or have had tubal ligation at least one year prior to Screening, or have had a total hysterectomy or bilateral salpingo-oophorectomy.
* Female Participants of child-bearing potential who are sexually active must consent to use an effective method of contraception as determined by the site investigator (i.e. oral hormonal contraceptives, patch hormonal contraceptives, vaginal ring, intrauterine devices, surgical hysterectomy, vasectomy, tubal ligation, or true abstinence) from the period following the signing of the informed consent through 12 weeks after the last dose of study drug.

Exclusion Criteria:

* Hypocalcemia or hypercalcemia, defined as serum calcium levels outside the age-adjusted normal limits and deemed as clinically significant in the opinion of the investigator.
* Vitamin D deficiency (25OH D3 < 20ng/ml); if Vitamin D is low at screening, substitution is allowed and recompensation has to be confirmed before treatment start by normalized levels of Vitamin D (25OH D3 ≥ 20ng/ml)
* Serum intact parathyroid hormone (iPTH) >2.5-fold the upper limit of normal (ULN)
* Severe renal insufficiency with a Glomerular filtration rate (eGFR) <30 at screening
* Treatment with oral phosphate and / or active vitamin D analogues in addition to Burosumab treatment. (In order to ensure appropriate patient care and preclude any harm due to deficient supply, required supplementation with oral phosphate salts and/or active vitamin D analogues at screening can be continued during the run-in phase but has to be stopped before Baseline and Initiation of treatment with Burosumab.)
* Treatment with bisphosphates or Denosumab within the last 6 months
* Treatment with Teriparatide within the last 3 months
* Intake of calcimimetics within 30 days before screening
* Patients with known hypersensitivity to Burosumab and the active substances of any of the excipients of Burosumab
* Presence of a concurrent disease or condition that would interfere with study participation or affect safety in the opinion of the investigator
* Use of any investigational product other than Burosumab or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Effect of Burosumab treatment on attaining serum phosphorus levels within the normal range in adults with XLH | 48 weeks
  Proportion of subjects attaining a serum phosphorus concentration within the normal range

SECONDARY OUTCOMES:
Change in chari rise test completion time | 48 weeks
  Change in chair rise test completion time from baseline to end of study visit
Change in 6-Minute-Walk test | 48 weeks
  Change in 6-Minute-Walk test distance from baseline to end of study visit
Change in timed up-and down stairs completion time | 48 weeks
  Change in timed up-and down stairs completion time from baseline to end of study visit
Normalization of TmP/GFR | 48 weeks
  Normalization of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate (TmP/GFR), proportion of subjects achieving normal values
Activity tracking | 48 weeks
  Activity tracking using 'Actibelt', to delineate total hours of physical activity per week

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Seefried, MD, Principal Investigator — University Hospital Wuerzburg
Locations (1):
- Clinical Trial Unit, Orthopedic Department, Wuerzburg University, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No
Only aggregated, analyzed participant data will be shared